CLINICAL TRIAL: NCT01087398
Title: Hematopoietic Stem Cell Transplantation for Malignant Infantile Osteopetrosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HORCSCT-0905
Record Dates: First submitted 2010-03-13; First posted 2010-03-16 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Osteopetrosis
Keywords: Osteopetrosis; HSCT
MeSH Terms: conditions — Osteopetrosis | interventions — Busulfan; Cyclophosphamide; thymoglobulin; fludarabine; Transplantation Conditioning; Neoadjuvant Therapy; Stem Cell Transplantation; Cyclosporine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental)
  Interventions: Drug: Busulfan, Cyclophosphamide, Thymoglobulin, Fludarabine (Conditioning regimen); Procedure: Stem Cell Transplantation; Drug: Cyclosporin, Methotrexate (GVHD prophylaxis)

INTERVENTIONS:
Drug: Busulfan, Cyclophosphamide, Thymoglobulin, Fludarabine (Conditioning regimen) — For sibling full match:
  * Busulfan 16 mg/kg >5year - 20 mg/kg <5year po
  * Cyclophosphamide 200 mg/kg iv
  For other related full match, sibling or other related with one antigen mismatch and umbilical cord blood:
  * Busulfan 16 mg/kg >5year - 20 mg/kg <5year po
  * Cyclophosphamide 200 mg/kg iv
  * ATG rabbit (Thymoglobulin) 10 mg/kg or ATG horse (Atgam) 40 mg/kg
  For haploidentical:
  * Busulfan 16 mg/kg >5year - 20 mg/kg <5year po
  * Cyclophosphamide 200 mg/kg iv
  * Fludarabine 160 mg/m^2
  Other Names: Systemic chemotherapy
Procedure: Stem Cell Transplantation — Patients undergoing Hematopoietic Stem Cell Transplantation from one of below source:
  1. Sibling full match
  2. Other related full match
  3. Sibling or other related with 1 mismatch antigen
  4. Cord Blood
  5. Haploidentical
  Other Names: HSCT
Drug: Cyclosporin, Methotrexate (GVHD prophylaxis) — * Cyclosporin A 1.5 mg/kg/day iv from -2, then 3 mg/kg/day iv (from +7 in PBSCT and +11 in BMT or UCBT) then 9 mg/kg/day po
  * 10 mg/m^2 iv day +1 then 6 mg/m^ iv day +3 and +6 (Not for UCBT)
  Other Names: Graft-versus-host disease (GVHD) prophylaxis

SUMMARY:
The purpose of this study is to evaluate the efficacy and side effects of donor hematopoietic cells using chemotherapy regimen without total-body irradiation in children undergoing a hematopoietic stem cell transplant for Malignant infantile osteopetrosis. The blood stem cells will be derived from either related donor or unrelated umbilical cord blood or haploidentical donor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Osteopetrosis confirm by bone biopsy and radiographic imaging
* Age up to 5 year old

Exclusion Criteria:

* Carbonic Anhydrase II (CAII) deficiency osteopetrosis variant
* Creatinine clearance ≤ 40ml/min/1.73m^2 or RTA
* Bilirubin ≥ 3mg/dL
* SGPT ≥ 500 U/L
* Current severe infection
* Evidence of CNS involvement
* Morbidity such as blindness or deafness

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival and Progressive Free Survival in patient with infantile Osteopetrosis who receive allogeneic HSCT | 1 year

SECONDARY OUTCOMES:
One year overall survival after allogeneic HSCT | 1 year
One year Progressive Free Survival after allogeneic HSCT | 1 year
Transplantation Related Mortality (TRM) after allogeneic HSCT | 1 year
Acute and chronic GVHD rate after allogeneic HSCT | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amir Ali Hamidieh, MD, Principal Investigator — Hematology-Oncology and SCT Research Center
Locations (1):
- Hematology-Oncology & SCT Research Center, Tehran, Tehran Province, Iran